CLINICAL TRIAL: NCT04028466
Title: Effectiveness of Vonoprazan vs Omeprazole as Empiric Therapy for Gastroesophageal Reflux Disease (GERD) Patients Without Alarm Features in a Primary Care Setting: A Pragmatic, Randomized, Single Blind Study
Brief Title: Effectiveness of Vonoprazan vs Omeprazole as Empiric Therapy for Gastroesophageal Reflux Disease (GERD) Patients Without Alarm Features
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Budget for the study was withdrawn and discontinued
Sponsor: St. Luke's Medical Center, Philippines (Other)
Responsible Party: Principal Investigator, Nicodemus Ong, Fellow and Principal Investigator, Institute of Digestlve and Liver Diseases, St. Luke's Medical Center, Philippines
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RP 19-007
Record Dates: First submitted 2019-07-06; First posted 2019-07-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: GERD; Gastro Esophageal Reflux
Keywords: GERD; gastro esophageal reflux; proton pump inhibitor; Potassium-Competitive Acid Blocker; H(+)-K(+)-Exchanging ATPase; Randomized Controlled Trial
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Omeprazole

STUDY DESIGN:
Intervention Model Description: Pragmatic, Randomized, Single Blind Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Randomized, Single Blind Study. Only primary investigators are blinded. the primary investigator also are the outcome assessors
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vonoprazan (Experimental): Patients will be randomized to receiving vonoprazan, which will be taken 30 minutes before the first meal of the day for 14 days
  Interventions: Drug: Vonoprazan
- Omeprazole (Active Comparator): Patients will be randomized to receiving omeprazole, which will be taken 30 minutes before the first meal of the day for 14 days
  Interventions: Drug: Omeprazole

INTERVENTIONS:
Drug: Vonoprazan — Patients will be randomized to receiving vonoprazan 20mg tablet or omeprazole 40mg capsule, either of which will be taken 30 minutes before the first meal of the day for 14 days
  Other Names: Investigational Arm
  Arms: Vonoprazan
Drug: Omeprazole — Patients will be randomized to receving vonoprazan 20mg tablet or omeprazole 40mg capsule, either of which will be taken 30 minutes before the first meal of the day for 14 days
  Other Names: Control Arm
  Arms: Omeprazole

SUMMARY:
Gastroesophageal reflux disease is a commonly encountered disorder in daily practice. Proton pump inhibitor therapy has been the cornerstone of treatment for decades. Although it has been proven to be highly effective, there is still room for improvement. A local study showed that only 57.3% of subjects are asymptomatic after 4 weeks treatment with rabeprazole. Recently a new drug was developed with better absorption, higher bioavailability, more sustained increased pH in the stomach and more targeted action to the H-K ATPase pump. Vonoprazan, belongs to a new class of acid suppressant medications, the potassium-competitive acid blocker (P-CAB). Vonoprazan has been studied and used successfully in Japan for H pylori eradication therapy, GERD, gastric and duodenal ulcers with favorable safety profile. However, to the author's knowledge, no study yet exists comparing vonoprazan to a proton pump inhibitor in the treatment of GERD outside Japan. This study aims to determine whether vonoprazan is superior to omeprazole in relieving symptoms in treatment-naïve adult patients with GERD.

DETAILED DESCRIPTION:
Gastroesophageal Reflux Disease (GERD) is globally defined as a condition that develops when the reflux of stomach contents causes troublesome symptoms and/or complications. The Philippine Clinical Practice Guideline on the Diagnosis and Treatment of GERD defined is as a condition resulting from recurrent backflow of gastric contents into the esophagus and adjacent structures causing troublesome symptoms and/or tissue injury. It is a commonly encountered disorder in the clinics and daily practice. A clinical diagnosis of GERD is acceptable with typical symptoms of acid regurgitation and/or heartburn is present. The Philippine guidelines state that empiric therapy can be started in GERD patients without alarm features and don't require further laboratory exam or workup. The guideline recommends standard dose proton pump inhibitor (PPI) therapy once daily for 8 weeks as cornerstone for treatment.

Proton pump inhibitor (PPI) therapy has been used as first line therapy of reflux symptoms for more than a decade. Even though it has been proven to be highly effective for reflux symptoms, there are still unaddressed issues. A local study by Lontok et al in 2013 evaluated response of GERD patients to rabeprazole 20mg once daily using a locally validated Frequency Scale of Symptoms of GERD (FSSG) in a primary care setting. Their study showed that a 4 week rabeprazole therapy resulting in complete resolution of individual symptoms ranging from 81.9-90.3%, with only 57.3% of all subjects being completely asymptomatic at the end of treatment. Proton pump inhibitors also have unmet issues needing improvement. PPIs usually takes 5 days for their maximal effect. Because of their slow onset of action, a significant number of patients are not sufficiently relieved after the first dose of PPI. Approximately half of patients still have symptoms after 3 days of treatment. PPIs are influenced by the cytochrome P450 (CYP) 2C19 polymorphism, with rapid metabolizers having the lowest intragastric pH compared with slow metabolizers. PPIs are also not sufficiently effective in controlling nocturnal heartburn symptoms because overnight recovery of gastric acid is frequently seen, therefore causing loss of sleep and health-related reductions in quality of life.

Recently, a new drug that promises better pharmacokinetic and pharmacodynamics properties was developed. Its use has been mostly in Japan for the past 2 years. Vonoprazan, is a novel, potassium-competitive acid blocker (P-CAB) that binds and inhibits H-K ATPase, the final step in acid secretion from the parietal cells of the stomach. It can inhibit the proton pump in both acidic and neutral environments with high affinity. The drug is retained for a long time inside the parietal cells and can inhibit H-K ATPase that is activated by further stimulation of acid secretion. Vonoprazan offers the advantage of not being required to be taken before meals, compared to conventional PPIs where 30 minutes before a meal is required, and is unaffected by the CYP2C19 polymorphism. Vonoprazan is also effectively absorbed and quickly accumulates in parietal cells, therefore, acid inhibition is more pronounced after the first dose of vonoprazan, compared to conventional PPIs where it usually takes 3-5 days for maximal effect. Vonoprazan is therefore, a stronger acid blocker that has rapid, stable and longer-lasting effects. Of the author's knowledge only 2 large scale randomized controlled trial have been done with vonoprazan, both these studies were done in Japan and focus only on those with erosive esophagitis. Vonoprazan has been showed to be effective and noninferior to lansoprazole for curing erosive esophagitis, as well as PPI resistant erosive esophagitis, with healing rates more pronounced for Grade C and D erosive esophagitis. Other studies on the use of vonoprazan for GERD have been done only in Japan, and comprised of noninferiority and small retrospective open label trials.

When vonoprazan is used for short term acid suppression, there are no problematic side effects. Treatment emergent adverse events irrespective of causal relationship to study medication are nasopharyngitis, diarrhea, constipation, upper respiratory infection, fall, gastroenteritis and eczema. Most of these treatment emergent adverse events were classified as mild in intensity. Studies are ongoing in Japan to assess the long term safety and efficacy of vonoprazan

. The Philippine Clinical Practice Guideline for GERD recommends locally-validated standardized questionnaire to assess treatment response to GERD. Commonly used questionnaires in the Philippines are the Frequency Scale for Severity of GERD (FSSG) and the Gastroesophageal Reflux Disease Questionnaire (GERDQ); both have undergone local validation studies. FSSG has been shown to correlate with endoscopic severity of GERD and assess response to proton pump inhibitor therapy.2 The FSSG comprises 12 questions where patients would rate individual symptoms as never (0% of the time), occasionally (around 30% of the time), sometimes (50%), often (70%) or always (100%). GERD is diagnosed if the score is more than 8, with sensitivity of 62%, specificity of 59% and accuracy of 60% for endoscopic diagnosis of esophagitis.

Vonoprazan was just recently introduced to the Philippine market recently. Whether or not this drug may replace conventional PPIs as first line therapy remains to be determined. This study aims to determine whether vonoprazan is superior to omeprazole in treating treatment-naïve adult patients with GERD. Data from this study will help formulate policies and recommendations on the treatment of GERD, as well as formulate new treatment strategies for patients with GERD.

ELIGIBILITY:
Inclusion Criteria:

* All Adult patients with clinically diagnosed with Gastroesophageal Reflux Disease (GERD) without alarm features (heartburn and acid regurgitation)
* Age more than 18 years at the time of written consent
* Those who provide written consent with their own free will
* Both treatment naïve and treatment experienced patients will be included. Treatment experienced patients should not be taking any proton pump inhibitors for 2 weeks to allow for washout period.

Exclusion Criteria:

* Patients that have alarm features as defined by the Philippines Guidelines for GERD (dysphagia, odynophagia, weight loss, anemia, hematemesis, family history of esophageal adenocarcinoma, nocturnal choking, abdominal mass, recurrent/frequent vomiting, chest pain)
* Patients with atypical GERD symptoms (cough, laryngitis, chest pain, etc.)
* Patients already taking proton pump inhibitors for the past 2 weeks
* Patients who scored less than 8 on the FSSG questionnaire
* Patients who have undergone gastroesophageal surgery
* Patients who are poorly compliant to medications
* allergy to PPI or vonoprazan
* With serious comorbidities, such as but not limited to: heart failure, renal failure, malignancy or hepatic failure
* Pregnant, breastfeeding or possibly pregnant
* Patients that would not provide consent
* Patients who are unable to complete the FSSG Questionnaire independently
* Patients who are unable to follow up at designated periods
* Patients taking rilpivirine or atazanavir.
* Patients with elevated baseline liver function tests (more than twice the upper limit of normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Proportion of asymptomatic patients at Day 3 | day 3 of therapy
  Asymptomatic patients is defined as a patient being free of symptoms of heartburn or acid regurgitation according to FSSG questionnaire (score <8) Expressed in percentage
Proportion of asymptomatic patients at Day 7 | day 7 of therapy
  Asymptomatic patients is defined as a patient being free of symptoms of heartburn or acid regurgitation according to FSSG questionnaire (score <8) Expressed in percentage
Proportion of asymptomatic patients at Day 14 | day 14 of therapy
  Asymptomatic patients is defined as a patient being free of symptoms of heartburn or acid regurgitation according to FSSG questionnaire (score <8) Expressed in percentage

SECONDARY OUTCOMES:
Proportion of partial responders at Day 3 | day 3 of therapy
  Partial responder are patients who still have GERD symptoms, but with partial improvement on reevaluation using the FSSG questionnaire; patients with at least 50% reduction from the baseline FSSG score Expressed in percentage
Proportion of partial responders at Day 7 | day 7 of therapy
  Partial responder are patients who still have GERD symptoms, but with partial improvement on reevaluation using the FSSG questionnaire; patients with at least 50% reduction from the baseline FSSG score Expressed in percentage
Proportion of partial responders at Day 14 | day 14 of therapy
  Partial responder are patients who still have GERD symptoms, but with partial improvement on reevaluation using the FSSG questionnaire; patients with at least 50% reduction from the baseline FSSG score Expressed in percentage
Proportion of nonresponders at Day 14 | day 14 of therapy
  Nonresponders are patients who reported no significant improvement in symptoms with treatment; patients with less than 50% reduction from the baseline FSSG score Expressed in percentage
Percent change in the symptom score from baseline (Vonoprazan Group) - Day 3 | day 3 of therapy
  Difference in the symptom score from baseline using the FSSG questionnaire at each time point within Vonoprazan and omeprazole group; expressed in percentage
Percent change in the symptom score from baseline (Vonoprazan Group) - Day 7 | day 7 of therapy
  Difference in the symptom score from baseline using the FSSG questionnaire at each time point within Vonoprazan and omeprazole group; expressed in percentage
Percent change in the symptom score from baseline (Vonoprazan Group) - Day 14 | day 14 of therapy
  Difference in the symptom score from baseline using the FSSG questionnaire at each time point within Vonoprazan and omeprazole group; expressed in percentage
Difference in percent change in the symptom score (between groups) | day 3, 7, and 14 of therapy
  Difference in the percent change of the FSSG score between groups will be analyzed using independent T test or Mann-Whitney U test between vonoprazan and omeprazole groups at one point in time
Number of Patients with Adverse Effects | Day 14 of therapy
  Safety and frequency of adverse effects experienced by patients (nasopharyngitis, diarrhea, constipation, upper respiratory tract infection, gastroenteritis, eczema/allergy, hypergastrinemia)

CONTACTS AND LOCATIONS:
Overall Officials: Nicodemus L Ong, MD, Principal Investigator — Institute of Digestive and Liver Diseases, St. Luke's Medical Center, Quezon City; Sherrie Isabel Q De Ocampo, MD, Principal Investigator — Institute of Digestive and Liver Diseases, St. Luke's Medical Center, Quezon City
Locations (1):
- St. Luke's Medical Center, Quezon City, National Capital Region, Philippines

IPD SHARING:
Plan to Share IPD: Undecided
Approval from the Institutional review board should be secured before IPD will be made available

REFERENCES:
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Cederberg C, Lind T, Rohss K, Olbe L. Comparison of once-daily intravenous and oral omeprazole on pentagastrin-stimulated acid secretion in duodenal ulcer patients. Digestion. 1992;53(3-4):171-8. doi: 10.1159/000200992. PMID 1291405
- [Background] Dammann HG, Burkhardt F. Pantoprazole versus omeprazole: influence on meal-stimulated gastric acid secretion. Eur J Gastroenterol Hepatol. 1999 Nov;11(11):1277-82. PMID 10563540
- [Background] Bytzer P, Morocutti A, Kennerly P, Ravic M, Miller N; ROSE Trial Investigators. Effect of rabeprazole and omeprazole on the onset of gastro-oesophageal reflux disease symptom relief during the first seven days of treatment. Scand J Gastroenterol. 2006 Oct;41(10):1132-40. doi: 10.1080/00365520600615781. PMID 16990197
- [Background] Peura DA, Riff DS, Snoddy AM, Fennerty MB. Clinical trial: lansoprazole 15 or 30 mg once daily vs. placebo for treatment of frequent nighttime heartburn in self-treating subjects. Aliment Pharmacol Ther. 2009 Sep 1;30(5):459-68. doi: 10.1111/j.1365-2036.2009.04064.x. Epub 2009 Jun 11. PMID 19523177
- [Background] Chong E, Ensom MH. Pharmacogenetics of the proton pump inhibitors: a systematic review. Pharmacotherapy. 2003 Apr;23(4):460-71. doi: 10.1592/phco.23.4.460.32128. PMID 12680476
- [Background] Furuta T, Shirai N, Sugimoto M, Nakamura A, Hishida A, Ishizaki T. Influence of CYP2C19 pharmacogenetic polymorphism on proton pump inhibitor-based therapies. Drug Metab Pharmacokinet. 2005 Jun;20(3):153-67. doi: 10.2133/dmpk.20.153. PMID 15988117
- [Background] Katz PO, Castell DO, Chen Y, Andersson T, Sostek MB. Intragastric acid suppression and pharmacokinetics of twice-daily esomeprazole: a randomized, three-way crossover study. Aliment Pharmacol Ther. 2004 Aug 15;20(4):399-406. doi: 10.1111/j.1365-2036.2004.02079.x. PMID 15298633
- [Background] Johnson DA, Katz PO. Nocturnal gastroesophageal reflux disease: issues, implications, and management strategies. Rev Gastroenterol Disord. 2008 Spring;8(2):98-108. PMID 18641592
- [Background] Fass R, Chey WD, Zakko SF, Andhivarothai N, Palmer RN, Perez MC, Atkinson SN. Clinical trial: the effects of the proton pump inhibitor dexlansoprazole MR on daytime and nighttime heartburn in patients with non-erosive reflux disease. Aliment Pharmacol Ther. 2009 Jun 15;29(12):1261-72. doi: 10.1111/j.1365-2036.2009.04013.x. Epub 2009 Apr 8. PMID 19392864
- [Background] Kusano M, Shimoyama Y, Sugimoto S, Kawamura O, Maeda M, Minashi K, Kuribayashi S, Higuchi T, Zai H, Ino K, Horikoshi T, Sugiyama T, Toki M, Ohwada T, Mori M. Development and evaluation of FSSG: frequency scale for the symptoms of GERD. J Gastroenterol. 2004 Sep;39(9):888-91. doi: 10.1007/s00535-004-1417-7. PMID 15565409
- [Result] Oshima T, Miwa H. Potent Potassium-competitive Acid Blockers: A New Era for the Treatment of Acid-related Diseases. J Neurogastroenterol Motil. 2018 Jul 30;24(3):334-344. doi: 10.5056/jnm18029. PMID 29739175
- [Result] Ashida K, Sakurai Y, Hori T, Kudou K, Nishimura A, Hiramatsu N, Umegaki E, Iwakiri K. Randomised clinical trial: vonoprazan, a novel potassium-competitive acid blocker, vs. lansoprazole for the healing of erosive oesophagitis. Aliment Pharmacol Ther. 2016 Jan;43(2):240-51. doi: 10.1111/apt.13461. Epub 2015 Nov 11. PMID 26559637
- [Result] Iwakiri K, Sakurai Y, Shiino M, Okamoto H, Kudou K, Nishimura A, Hiramatsu N, Umegaki E, Ashida K. A randomized, double-blind study to evaluate the acid-inhibitory effect of vonoprazan (20 mg and 40 mg) in patients with proton-pump inhibitor-resistant erosive esophagitis. Therap Adv Gastroenterol. 2017 Jun;10(6):439-451. doi: 10.1177/1756283X17705329. Epub 2017 Apr 25. PMID 28567114
- [Result] Shinozaki S, Osawa H, Hayashi Y, Sakamoto H, Kobayashi Y, Lefor AK, Yamamoto H. Vonoprazan 10 mg daily is effective for the treatment of patients with proton pump inhibitor-resistant gastroesophageal reflux disease. Biomed Rep. 2017 Sep;7(3):231-235. doi: 10.3892/br.2017.947. Epub 2017 Jul 20. PMID 28894571
- [Result] Kinoshita Y, Sakurai Y, Shiino M, Kudou K, Nishimura A, Miyagi T, Iwakiri K, Umegaki E, Ashida K. Evaluation of the Efficacy and Safety of Vonoprazan in Patients with Nonerosive Gastroesophageal Reflux Disease: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study. Curr Ther Res Clin Exp. 2016 Dec 21;81-82:1-7. doi: 10.1016/j.curtheres.2016.12.001. eCollection 2016. PMID 28119763
- [Result] Mori H, Suzuki H. Role of Acid Suppression in Acid-related Diseases: Proton Pump Inhibitor and Potassium-competitive Acid Blocker. J Neurogastroenterol Motil. 2019 Jan 31;25(1):6-14. doi: 10.5056/jnm18139. PMID 30504527

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT04028466/Prot_SAP_000.pdf